CLINICAL TRIAL: NCT00522600
Title: Evaluation of Eye Drop Administration in Glaucoma Patients
Brief Title: Eye Drop Use in Glaucoma Patients Through Patient Surveys and Video Observations
Status: Completed | Type: Observational
Sponsor: Robin, Alan L., M.D. (Individual)
Collaborators: Alcon Research (Industry)
Responsible Party: Jennifer L. Stone, OD, Glaucoma Specialists
Other Study IDs: SI0717
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Glaucoma; Dry Eye Syndrome; Conjunctivitis
Keywords: eyedrops; compliance; glaucoma medications; adherence
MeSH Terms: conditions — Glaucoma; Dry Eye Syndromes; Conjunctivitis; Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be used to evaluate how patients put eye drops in their eyes and any problems that may arise from this activity. The information gathered will help identify common problems patients are having with putting in their eye medications. Then doctors can be better informed about the issues and provide better advice to their patients to overcome these problems.

DETAILED DESCRIPTION:
Approximately 100 patients will take part in a one time procedure and survey as part of this project. After appropriate consent patients are asked to complete a short 2 page survey about themselves and their eye drops. Then a video recording will be made of the patient instilling eye drops in their habitual manner. The eye drops used will be sterile saline placed in either Travatan-like or Systane bottles to simulate the corresponding prescribed medication. The videos will be graded for instillation technique and combined with scoring of survey answers.

Patients will be asked to instill the drops to their left eye with their dominant hand as we expect this to be most difficult. Patients with severe (>20/200) vision loss will instill drops into their better seeing eye.

ELIGIBILITY:
Inclusion Criteria:

* Currently using topical glaucoma medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 173 subjects enrolled and 222 video recordings were made. Ages ranged from 21-94 years old (mean:67 yrs) and subjects were 55% female and 70% caucasian.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-02; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Stone, OD, Principal Investigator — Alan L Robin MD PA; Alan L Robin, MD, Study Director — Alan L Robin MD PA
Locations (1):
- ALan L Robin MD PA, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Stone JL, Robin AL, Novack GD, Covert DW, Cagle GD. An objective evaluation of eyedrop instillation in patients with glaucoma. Arch Ophthalmol. 2009 Jun;127(6):732-6. doi: 10.1001/archophthalmol.2009.96. PMID 19506189